CLINICAL TRIAL: NCT02109549
Title: Influence of Metformin Use on Treatment Outcome in NSCLC Patients
Brief Title: Influence of the Use of the Diabetic Drug Metformin on the Overall Survival and Treatment-related Toxicity in Advanced Stage Non-small Cell Lung Cancer Patients.
Acronym: Metformin
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastro Clinic, The Netherlands (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Other Study IDs: Metformin NSCLC
Record Dates: First submitted 2014-03-26; First posted 2014-04-10 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Diabetes and metformin: Patients with diabetes mellitus treated with metformin only.
- Insulin-diabetes without metformin: Patients with insulin-dependent diabetes mellitus not treated with metformin
- Controlgroup: The remaining patients serve as control group.

SUMMARY:
There are preliminary data suggesting that patients suffering from non-insulin-dependent diabetes mellitus, treated with metformin, have improved local tumor control. A reduction in the tumor's hypoxia may be responsible for this phenomenon.

Therefore, the aim of this study is to test the hypothesis in three cohorts of patients suffering from advanced stage non-small cell lung cancer and all undergoing concurrent radiochemotherapy: 1. Patients with diabetes mellitus treated with metformin only; 2. Patients with insulin-dependent diabetes mellitus not treated with metformin; 3. The remaining patients serving as controls. Furthermore, tumor and treatment-related parameters will be correlated with overall survival and morbidity.

DETAILED DESCRIPTION:
There are preliminary clinical and preclinical data suggesting that patients suffering from non-insulin-dependent diabetes mellitus, treated with metformin, have improved local tumor control. The reduction in oxygen consumption of tumor cells and thus a relative reduction in the tumor's hypoxia may be responsible for this.

Non-small cell lung cancer is the most frequent solid tumor in many Western countries and the number one cause of cancer-related death. Even though the introduction of concurrent chemoradiotherapy has improved local tumor control and thus overall survival, 5-year overall survival is still as low as 14%. Furthermore, many patients are not eligible to undergo concurrent treatment thus reducing their chances to defeat this disease. Additionally, concurrent chemoradiotherapy is associated with increased toxicity compared to sequential treatment. Therefore, alternative additives improving the effect of radiotherapy without increasing toxicity to an unbearable level are searched for. One possible pharmaceutical is metformin; many patients have been using it in the past without evident increased toxicity, it is cheap, and widely available.

Thus, the aim of this study is to test the hypothesis that metformin increases overall survival without enhancing treatment-related toxicity. For this means, in three cohorts of patients suffering from advanced stage non-small cell lung cancer and all undergoing concurrent radiochemotherapy: 1. Patients with diabetes mellitus treated with metformin only; 2. Patients with insulin-dependent diabetes mellitus not treated with metformin; 3. The remaining patients serving as controls. Using Kaplan-Meier statistics as well as uni- and multivariate analysis, the overall survival and toxicity of these cohorts will be compared. Other potentially confounding factors will be tested as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

Advanced non-small cell lung cancer patients undergoing primary concurrent radiochemotherapy; patients treated with metformin or insulin will be analyzed as separate cohorts.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced stage non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Assessment of metformin use | 2 years after radiotherapy
  Assessment of metformin use (in patients with diabetes mellitus) on overall survival in advanced stage NSCLC patients undergoing radiochemotherapy.
Assessment of insulin use | 2 years after radiotherapy
  Assessment of insulin use (in patients with diabetes mellitus) on overall survival in advanced stage NSCLC patients undergoing radiochemotherapy.

SECONDARY OUTCOMES:
Overall assessment of overall survival and toxicity factors | 2 years after radiotherapy
  Composite outcome measure:
  Assessment of factors influencing overall survival and toxicity:
  Age Gender Performance status WHO TNM stage Histology Delivered radiation dose Total gross tumor volume Total planning target volume

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands; Esther Troost, Study Chair — Maastro Clinic, The Netherlands; José Belderbos, Principal Investigator — NKI Amsterdam; Edith Dieleman, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (3):
- Netherlands (3):
  - The Netherlands Cancer Institute (NKI), Amsterdam
  - AMC, Amsterdam
  - MAASTRO clinic, Maastricht